CLINICAL TRIAL: NCT02476604
Title: Seton Hill University--Personal Empowerment Program
Acronym: SHU-PEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Seton Hill University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 375278-3
Record Dates: First submitted 2015-06-09; First posted 2015-06-19 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular Diseases
Keywords: prevention; adult; student
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Messaging (Experimental): Subjects randomized to the intervention arm will receive health coaching and electronic messages at the rate of up to six times per week over an 8 week period.
  Interventions: Behavioral: health coaching and electronic messaging
- Control (No Intervention): Subjects randomized to the control arm will undergo all of the same measurements for baseline and follow up data but will not receive the intervention of health coaching and electronic messaging.

INTERVENTIONS:
Behavioral: health coaching and electronic messaging — Using using an iPAD or notebook PC, students will receive electronic messaging aimed at encouraging adherence to behavioral goals previously set via discussions with the health coaches. The messages will be received 3 to 6 times per week for the 8 week intervention period.
  Arms: Electronic Messaging

SUMMARY:
It is widely acknowledged that cardiovascular disease prevention requires intervention as early in the human lifespan as practical. A window of opportunity presents in early adulthood when students gain independence as young adults attending university. In a three-phase investigation, this study will evaluate the behavioral patterns of university students in the domains of diet, exercise, stress management, smoking and sleep (phase 1). Informed with information from phase 1, a pilot study (phase 2) will test the feasibility of performing an intervention in university students consisting of an 8-week period during which the students will receive up to six text messages (by phone or iPad) per week, tailored to address the behavioral issues that the student has identified as needing improvement and for which the student has indicated a desire to make change. Using lessons learned in phase 2, a randomized, controlled trial of the 8 week intervention (phase 3) will compare intervention subjects with controls for outcomes of behavior change, measures of anthropometric data, and serum markers of cardiovascular risk to test the impact of the intervention

DETAILED DESCRIPTION:
This proposal aims to study the issues of health behaviors in the domains of diet, exercise, stress, and sleep. We aim to improve health behaviors in these domains by evaluating lifestyle choices and communication preferences with a three phase investigation. Phase 1 has the specific objective of lifestyle assessment. Phase 1 will evaluate dietary habits and choices, exercise practices, perceived stress levels, and quantity and timing of sleep utilizing a web-based health survey. The web-based survey tool will populate a secure research database. The data will include demographic information, anthropometric data, actigraphic data to measure exercise levels and sleep time, and laboratory studies that measure glucose metabolism, lipids, and other laboratory markers for cardiovascular risk assessment.

Phase 2 constitutes a pilot study in a limited number of university students to determine the feasibility of causing healthy behavior change with the use of electronic messaging to university students up to six times per week over 8 weeks. Experience from this feasibility study will inform the design of Phase 3.

Phase 3 will measure improvements in the lifestyle behaviors of students as a result of health coaching and electronic feedback messages over an 8 week period comparing their indices of health with a control group that does not receive the coaching and electronic feedback messages. Utilizing lessons learned from Phase 2, subjects randomized to an intervention arm but not subjects randomized to a control arm, will receive health coaching and electronic messages at the rate of up to six times per week over an 8 week period. Before and after this intervention period, measurements of lifestyle choices, anthropometrics, actigraphy for objective exercise and sleep patterns, and cardiac-relevant laboratory studies will be measured. Data from the intervention group will be compared with that of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Full time undergraduate student at Seton Hill University
* Ages 18 to 30 years
* Healthy

Exclusion Criteria:

* Part-time study (less than 12 semester hours of enrollment)
* Under 18 years or over 30 years of age
* Pregnant or planning to become pregnant during study
* Diagnosed eating disorder
* Diagnosed with chronic medical illness such as heart disease (including pacemaker placement), gastro-intestinal disease, diabetes, pulmonary disease
* Taking prescribed medication other than birth control pills or multivitamins on an ongoing basis
* Any condition that may preclude the ability to perform the requirements of the study (for example an orthopedic or neurological condition that prevents the accurate measurement of a subject's height).
* Persons with metal implants (plates, etc)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
A composite score for adherence to personal goals for Diet, Exercise, Stress Management and Expansion of Sleep Time. | 8 weeks
  Improvement will be determined by calculating a composite score for % achievement in adhering to goals set for Rate-Your-Plate Dietary Assessment, Exercise Minutes, Stress Reduction by Perceived Stress Scale and Total Sleep Time.

SECONDARY OUTCOMES:
Weight Management | 8 weeks
  BMI and % body fat changes
Lipid Profile | 8 weeks
  Change in chemical profile of lipid panel
Glucose Metabolism | 8 weeks
  Change in fasting glucose
Hemoglobin A1C | 8 weeks
  Change in hemoglobin A1C

CONTACTS AND LOCATIONS:
Overall Officials: Arn Eliasson, MD, Study Director — Walter Reed National Military Medical Center
Locations (2):
- United States (2):
  - Integrative Cardiac Health Project, Walter Reed National Military Medical Center, Bethesda, Maryland
  - Seton Hill University, Greensburg, Pennsylvania

REFERENCES:
- [Derived] Sandrick J, Tracy D, Eliasson A, Roth A, Bartel J, Simko M, Bowman T, Harouse-Bell K, Kashani M, Vernalis M. Effect of a Counseling Session Bolstered by Text Messaging on Self-Selected Health Behaviors in College Students: A Preliminary Randomized Controlled Trial. JMIR Mhealth Uhealth. 2017 May 17;5(5):e67. doi: 10.2196/mhealth.6638. PMID 28526664